CLINICAL TRIAL: NCT03701178
Title: One Year Clinical Evaluation of Milled BioHPP Polyetheretherketone (PEEK) Versus Zirconia Veneered Single Crowns (Randomized Controlled Clinical Trial-one-year Evaluation).
Brief Title: One Year Clinical Evaluation of Milled BioHPP (PEEK) Versus Zirconia Veneered Single Crowns (RCT-one-year Evaluation).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mustafa hassan, assistant lecturer , fixed prosthodontic department, faculty of dentistry ERU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-38
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Carious Tooth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zirconia veneered crowns (Active Comparator): we will use zirconia veneered single crowns as a control to evaluate the marginal integrity and fracture and patient satisfaction
  Interventions: Other: BioHPP PEEK
- milled BioHpp PEEK (Experimental): we will use milled BioHPP PEEK single crowns as a intervention to evaluate the marginal integrity and fracture and patient satisfaction
  Interventions: Other: BioHPP PEEK

INTERVENTIONS:
Other: BioHPP PEEK — milled BioHPP PEEK in a new material can be used as a dental restoration

SUMMARY:
All ceramic crowns are indicated in case of mild to moderate discoloration, restoration of traumatized or fractured teeth and abnormal tooth anatomy. Long term success of all ceramic crowns is affected by many factors. Fracture of the all ceramic crowns is the most repeated failure pattern and represents about 67% of total failures associated with this type of restoration through a period of 15 years of clinical performance.

Polyetheretherketone (PEEK) is a polymer that has many potentials uses in dentistry. Polyetheretherketone (PEEK) can be used to support fixed dental prostheses. However, information about physio mechanical characterization is still scarce.

DETAILED DESCRIPTION:
Polyetheretherketone (PEEK) is a synthetic, tooth colored polymeric material that has been used as a biomaterial in orthopedics for many years due to its lower Young's (elastic) modulus (3-4 GPa) being close to human bone. PEEK can be modified easily by incorporation of other materials. For example; incorporation of carbon fibers or glass fibers can increase the elastic modulus up to 18 GPa which becomes comparable to those of cortical bone and dentin so the polymer could exhibit good stress distribution . Moreover, tensile properties of PEEK are also analogous to those of bone, enamel and dentin making it a suitable restorative material as far as the mechanical properties are concerned.

BioHPP PEEK is 20% ceramic reinforced, semicrystalline, thermoplastic and radiolucent polymer for extreme durability especially for frameworks for fixed and removable dental prostheses. It has many advantages as low density, light weight, shock absorber, biocompatible and venerable with composite resin.

BioHPP PEEK can be fabricated via CAD/CAM technology by milling PEEK blanks. It is also can be pressed by using granular or pellet-shaped PEEK. Three-unit PEEK fixed partial denture manufactured via CAD-CAM has been suggested to have a higher fracture resistance than pressed granular- or pellet-shaped PEEK dentures.

The fracture resistance of the CAD/CAM milled PEEK fixed dentures is much higher than those of lithium disilicate glass-ceramic (950N), alumina (851N) , zirconia (981-1331N). The abrasive properties of PEEK are excellent. Despite of significantly low elastic moduli and hardness, abrasive resistance of PEEK is competitive with metallic alloys .

BioHPP PEEK can be used under resin composite as a coping material. Because the mechanical properties of PEEK are similar to those of dentin and enamel, PEEK could have an advantage over alloy and ceramic restorations . A variety of procedures have been suggested to condition the surface of PEEK in order to facilitate its bonding with resin composite crowns. For example, air abrasion with and without silica coating creates a more wettable surface. Etching with sulphuric acid creates a rough and chemically altered surface which enables it to bond more effectively with hydrophobic resin composites .

Due to these unique physical and mechanical properties, BioHPP PEEK is a promising material for dental application and it has been proposed for other prosthodontic applications such as fixed prostheses and removable prostheses .

ELIGIBILITY:
Inclusion Criteria:

* From 18-50 years old, be able to read and sign the informed consent document.
* Have no active periodontal or pulpal diseases, have teeth with good restorations
* Psychologically and physically able to withstand conventional dental procedures
* Patients with teeth problems indicated for single posterior crowns: (Badly decayed teeth / Teeth restored with large filling restorations / Endodontically treated teeth / Malformed teeth / Malposed teeth (Tilted, over-erupted, rotated, etc.) / Spacing between posterior teeth)
* Able to return for follow-up examinations and evaluation.

Exclusion Criteria:

* Patient less than 18 or more than 50 years
* Patient with active resistant periodontal diseases
* Patients with poor oral hygiene and uncooperative patients
* Pregnant women
* Patients in the growth stage with partially erupted teeth
* Psychiatric problems or unrealistic expectations
* Lack of opposing dentition in the area of interest

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
fracture | 1 year
  number of fracture

SECONDARY OUTCOMES:
marginal interity | 1 year
  marginal gap at the finish line

OTHER OUTCOMES:
patient satisfaction | 1 year
  patient satisfy from the color and anatomy of the restoration

CONTACTS AND LOCATIONS:
Overall Officials: abdelrahman M el sokkary, mastrer, Study Chair — researcher

IPD SHARING:
Plan to Share IPD: Undecided